CLINICAL TRIAL: NCT03625154
Title: Operative Versus Non Operative Management Outcomes of Isolated Lateral Malleolar Weber B Ankle Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Charles Moon, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro47932
Record Dates: First submitted 2018-06-28; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non operative control group (Active Comparator): Patients with negative gravity stress (non-operative treatment/observational control group)
  Interventions: Other: non operative management
- non operative experimental group (Active Comparator): Patients with positive gravity stress (medial clear space > 4 mm on initial injury pre-reduction x-rays, who undergo a reduction with closing of the medial clear space to <4mm. Plan for nonoperative treatment of all these patients with splint and subsequent walker boot.
  Interventions: Other: non operative management
- operative observational group (Active Comparator): Patients with positive gravity stress (medial clear space > 4 mm) who undergo a reduction with closing of the medial clear space to <4mm who declined non-operative treatment but agree to be observed. These patients will undergo ORIF (Open Reduction and Internal Fixation) with plates and screws and function as a second observation group
  Interventions: Procedure: ankle open reduction internal fixation

INTERVENTIONS:
Procedure: ankle open reduction internal fixation — Open Reduction and Internal Fixation with plates and screws
  Arms: operative observational group
Other: non operative management — closed reduction and splinting followed by progressive weight bearing
  Arms: non operative control group; non operative experimental group

SUMMARY:
The primary objective of this study is to determine the failure rate and difference in clinical outcomes between operative and non operative treatment of patients with Weber B lateral malleolus ankle fractures with medial clear space widening on gravity stress views. All patients presenting will be treated non operatively, and compared to an observational group comprised of patients with Weber B lateral malleolus ankle fractures without medial clear space widening, for which the standard of care is non operative management.

Patients who decline non operative management and elect to undergo operative open reduction internal fixation with plates and screws will comprise an operative observational cohort.

All patients will be followed for a total of 12 months from the time of injury. Clinical outcomes will be based on radiographic monitoring for ankle mortise congruency, as well as standardized SF-36 and AOFAS questionnaire scores.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* able to provide informed consent

Exclusion Criteria:

* pregnancy
* prisoners
* psychiatric conditions that prevent ability to provide informed consent or present barriers to follow up
* insulin dependent diabetics
* patients with prior musculoskeletal issues affecting the same extremity
* Patients cannot simultaneously be enrolled in any other studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-07-18 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
radiographic outcome of ankle congruency | 1 year
  measurement of medial clear space between medial malleolus and medial talar dome, measurement of tibiofibular overlap 1cm superior to the plafond, and measurement of superior clear space between the tibial plafond and the talar dome

SECONDARY OUTCOMES:
functional outcome by American Orthopedic Foot and Ankle Score (AOFAS) scoring system | 1 year
  total score 0-100, with 100 being the maximum best score. (pain (0-40 points), function (0-50 points) and alignment (0-10 points)
additional functional outcome by Short Form Survey (SF-36) Score scoring system | 1 year
  0 to 100 range, 100 being the best; subscores Physical functioning (0-10), Role limitations due to physical health (0-4), Role limitations due to emotional problems (0-3), Energy/fatigue (0-4)Emotional well-being (0-5), Social functioning (0-2), Pain (0-2), General Health 0-5
functional outcome by American Orthopedic Foot and Ankle Score (AOFAS) - Pain score | 1 year
  none, mild occasional, moderate daily, severe and almost always present
functional outcome by American Orthopedic Foot and Ankle Score (AOFAS) - function - activity limitations, support requirements | 1 year
  no limitations and no support, no limitation of daily activities but limitation of recreational activities, limited daily and recreational activities, or severe limitation of daily and recreational activities
functional outcome by American Orthopedic Foot and Ankle Score (AOFAS) - alignment | 1 year
  good plantigrade, midfoot well aligned; fair plamtigrade, some degree of midfoot malalignment, poor with nonplantigrade foot, severe malalignment